CLINICAL TRIAL: NCT05047120
Title: Hypnotic Cognitive Therapy During Inpatient Rehabilitation to Reduce Acute & Chronic SCI Pain: a Randomized Controlled Trial
Brief Title: Hypnotic Cognitive Therapy Reduce Acute & Chronic SCI Pain in Inpatient Rehabilitation
Acronym: HYPCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Craig H. Neilsen Foundation (Other)
Responsible Party: Principal Investigator, Amy Starosta, Assistant Professor, School of Medicine: Dept. of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009601
Record Dates: First submitted 2021-08-24; First posted 2021-09-16 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries; Pain, Chronic; Spinal Cord Injury, Acute
Keywords: Behavioral: Hypnotic Cognitive Therapy (HYPNOCT); spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypnosis Enhanced Cognitive Therapy (Experimental): This arm will receive 4 sessions of hypnosis enhanced cognitive therapy for pain. Subjects will receive recordings of sessions for practice between therapist sessions.
  Interventions: Behavioral: Hypnosis enhanced cognitive behavioral therapy
- Pain Education (Active Comparator): This arm will receive 4 sessions of spinal cord injury pain education. Subjects will receive pain education materials for review between therapist sessions.
  Interventions: Behavioral: Pain Education

INTERVENTIONS:
Behavioral: Hypnosis enhanced cognitive behavioral therapy — This therapy entails subjects being induced into a state of relaxation and the receiving cognitive behavioral therapy for pain associated with a new spinal cord injury.
  Other Names: HYPCT
  Arms: Hypnosis Enhanced Cognitive Therapy
Behavioral: Pain Education — This therapy entails subjects learning about the causes, mechanisms, and ways to reduce pain associated with a new spinal cord injury.
  Other Names: ED
  Arms: Pain Education

SUMMARY:
Chronic spinal cord injury (SCI) pain is complex and difficult to treat. For individuals with SCI, pain often begins early in the course of their SCI and continues longitudinally. Unfortunately, SCI-related pain is frequently not responsive to medical treatment and medical treatments that are available and commonly used, such as opioids, have negative side-effects and risk of addiction. Nonpharmacological (non-medication) interventions to reduce chronic pain show promise both for individuals with SCI as well as other chronic pain conditions. Research on psychological interventions for chronic pain over the past two decades has consistently found these interventions to be more effective than no treatment, standard care, pain education, or relaxation training alone. However, many of these interventions are designed and implemented in outpatient settings after chronic pain has already developed. The development of early, effective, and preventative interventions to reduce the development of chronic pain has the potential to vastly improve quality of life for individuals with SCI.

Having demonstrated the feasibility and acceptance of this treatment in an earlier study, the purpose of this randomized clinical trial is to compare the treatment of Hypnosis Enhanced Cognitive (HYPCT) therapy to Pain Education (ED) for reducing acute and chronic pain for individuals with new spinal cord injuries. The main goals of the study are to:

* Aim 1: Test the effectiveness of HYPCT during inpatient rehabilitation for SCI compared to a ED for reducing current pain intensity.
* Aim 2: Determine the post-intervention impact of HYPCT sessions compared to ED on average pain intensity.

Participants will be asked to:

* Complete 4 surveys over seven months
* Complete pre and post treatment pain assessments for each of 4 treatment/control sessions

Participants will be assigned to one of two groups for treatment and receive either:

* 4 Hypnotic Cognitive therapy sessions or
* 4 Pain Education sessions

DETAILED DESCRIPTION:
The purpose of this study is to see if a novel psychotherapy is helpful for reducing pain in patients who been recently diagnosed with a spinal cord injury (SCI). This therapy is an in-person hypnosis enhanced cognitive therapy designed to help people with a recent SCI cope with the pain that may come with that injury. Hypnosis enhanced cognitive therapy will be compared to pain education. Pain education is a semi-standard course which instructs patients with SCI about the types, causes, and usual treatments for pain associated with SCI. This study will be conducted with newly diagnosed patients completing their initial inpatient rehabilitation treatment at Harborview Medical Center in Seattle, WA.

Subjects who meet eligibility criteria and consent to take part in this study will be randomly assigned to one of two groups. One is hypnosis enhance cognitive therapy (HYPCT) group and the other is the pain education (ED) group. Subjects cannot choose which group to be in.

Hypnosis Enhance Cognitive Therapy Group:

Participants assigned to this group will work with a psychologist (PhD) who will provide them with HYPCT. There will be 4 therapy sessions spread out over the duration of the inpatient stay or at least weekly. Sessions will take place in patient hospital rooms and last approximately one hour. Patients will learn some new information and skills to better cope with pain. Sessions will include a brief hypnosis to help patients think about pain in ways that will reduce their experience of pain. During hypnosis, patients spend a lot of time relaxing and listening to the sound of the psychologist's voice. We will record these hypnosis exercises so that patients can listen to them in between sessions with the psychologist.

Pain Education Group:

Participants assigned to this group will work with a psychologist (PhD) who will provide them with ED. There will be 4 education sessions spread out over the duration of the inpatient stay or at least weekly. Sessions will take place in the patient hospital rooms and last approximately one hour. Patients will be educated about pain, including its causes, neurophysiology, nature, and impact. There may be both general pain information as well as information tailored to the SCI specific symptoms. These will be interactive and patients will discuss the content with the therapist. Patients may listen to audio recordings, review educational information and think about what they learned between sessions. Upon completing the study, everyone in the pain education group will be offered the 6 standardized hypnosis audio recordings provided to the HYPCT group. ED group will be asked to complete a survey one month after receiving the standard hypnosis recordings.

Both groups will be asked to complete a baseline survey asking about their demographics, health, and pain. A second survey will be completed after completion of the treatment sessions (HYPCT and ED), a survey will be completed 6 months after that, and then a final survey one month later (at approximately 7 months). The surveys will ask questions about the patient's pain, the treatment of their pain, mood, and sleep quality. A trained research assistant will administer the surveys in person during the rehabilitation hospital stay and by telephone after discharge. These surveys will each take 30-45 minutes. For both groups, before and after each session, patients will be asked about their pain levels and relief. This should take less than 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SCI at any level or severity
* currently admitted to IPR at Harborview Medical Center
* moderately intense pain
* evidences an ability to read and speak English

Exclusion Criteria:

* severe cognitive impairment
* presence or history of mental health problems that would require referral for more intensive treatment or complicate hypnotic treatment
* suicide attempt within the past 6 months
* current, active suicidal ideation, plan, or intent
* unable to provide informed consent.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
0-10 Numerical Rating Scale of Pain change score (Decrease in Pain following live Session with Therapist) | 2 times per week for 4 weeks
  0 - 10, self-reported rating of pain. Possible scores range from 0 (no pain) to 10 (pain as bad as you can imagine)
0-10 Numerical Rating Scale of Pain (Pain Relief following Practice Sessions) | 1 time per week for 4 weeks
  0 - 10, self-reported rating of pain. Possible scores range from 0 (no pain) to 10 (pain as bad as you can imagine)
Self-reported estimate of amount of time post therapy session that pain relief persists | 1 time per week for 4 weeks
  Minutes and/or hours after therapy that pain relief persists
Self-reported estimate of amount of time post practice session that pain relief persists | 1 time per week for 4 weeks
  Minutes and/or hours after practice session that pain relief persists
0-10 Numerical Rating Scale of Pain (Weekly average pain intensity) | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  0 - 10, self-reported rating of pain. Possible scores range from 0 (no pain) to 10 (pain as bad as you can imagine)

SECONDARY OUTCOMES:
PROMIS Pain Interference Short Form | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  The PROMIS Pain Interference measures the self-reported consequences of pain on relevant aspects of a person's life.
PHQ-9 | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  Patient Health Questionnaire is used to provisionally diagnose depression and grade severity of symptoms in general medical and mental health settings.
PROMIS Anxiety short form | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  PROMIS Anxiety short form is a 7-item measure that assesses the pure domain of anxiety in individuals.
PROMIS Sleep Disturbance | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  The PROMIS Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep.
Opioid Use from Electronic medical record review | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion)
  Medication and dosage
The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) | 1 time upon enrollment, time at 6 month Follow-up, 1 time at 7 month follow-up.
  The Tobacco, Alcohol, Prescription medications, and other Substance [TAPS] Tool consists of a 4-item screening for tobacco use, alcohol use, prescription medication misuse, and illicit substance use in the past year and brief assessment
0-10 Numerical Rating Scale of Pain (Pain Relief following Medication Administration) | 1 time per week for 4 weeks
  0-10 Numerical Rating Scale of Pain
Digit span (forward, backward, sequencing) (Working memory) | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  Measure ask subjects to count forward, backwards, and with different sequencing.

OTHER OUTCOMES:
Frequency of Independent Practice | 1 time per week for 4 weeks, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  Self-report of number of practice sessions
UW-CAP Short Form (Pain Catastrophizing) | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  The UW-CAP is intended measure an individual's level of pain catastrophizing.
Chronic Pain Acceptance Scale (Pain Acceptance) | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  Chronic Pain Acceptance Scale (Pain Acceptance) has been designed to measure acceptance of pain.
UW-PRSE Short Form (Pain Related Self-Efficacy) | 1 time upon enrollment, 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  The UW-PRSE is intended measure an individual's level of pain related self-efficacy.
Patient Global Impression of Improvement (PGI-I) | 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  The Patient Global Impression of Improvement (PGI-I) is an instrument designed to measure a patients interpretation of symptom changes following intervention.
Benefit, Satisfaction, and Willingness (BSW) | 1 time after 4 weeks (HYPCT/ED Completion), 1 time at 6 month Follow-up, 1 time at 7 month follow-up.
  The BSW is a useful tool to capture patients' global impressions of three key elements of treatment outcome: a perceived benefit, satisfaction with treatment, and the willingness to continue treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amy J Starosta, PhD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Starosta AJ, Bombardier CH, Kahlia F, Barber J, Accardi-Ravid MC, Wiechman SA, Crane DA, Jensen MP. Feasibility of Brief, Hypnotic Enhanced Cognitive Therapy for SCI-related Pain During Inpatient Rehabilitation. Arch Phys Med Rehabil. 2024 Jan;105(1):1-9. doi: 10.1016/j.apmr.2023.06.005. Epub 2023 Jun 25. PMID 37364685